CLINICAL TRIAL: NCT00506740
Title: A Randomized, Prospective, Parallel Group Study Comparing the Harmonic™ to Electrocautery in Abdominoplasties
Brief Title: Harmonic™ vs. Electrocautery in Abdominoplasties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CI-06-0002
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Skin and Fat Redundancy and Muscle Diastases
MeSH Terms: conditions — Diastasis, Muscle | interventions — Radionuclide Generators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrocautery (Active Comparator): Elesurgical instruments are used to cut and coagulate tissue using alternatig electric current focusing intense heat at the surgical site. In electrosurgery, the patient is included in the circuit and current enters the patient's body.
  Interventions: Device: Ultrasonic scalpel; Device: monopolar electrosurgery generator and tip

INTERVENTIONS:
Device: Ultrasonic scalpel — A surgical instrument that uses ultrasonic energy that allows both cutting and coagulating at the precise point of application.
  Other Names: 1) Sharp Curved Blade (HF105); 2) Generator (GEN04); 3) Hand Piece (HP054); Manufacturer: Ethicon Endo-Surgery, Inc., Cincinnati, OH.
Device: monopolar electrosurgery generator and tip

SUMMARY:
the objective of this study is to determine if the use of The Harmonic™ (an ultrasonic surgical instrument) in abdominolipectomy (tummy tuck)reduces volume and duration of wound drainage after surgery when compared to electrocautery.

DETAILED DESCRIPTION:
Abdominolipectomy is performed to correct abdominal skin and fat redundancy and muscle diastases. Persistent serous wound drainage and seromas are the most common complications in abdominolipectomy. The rate of serous fluid collection determines the time drains need to remain in place. Although suction drains reduce seroma formation, prolonged use can delay healing, cause injury, and increase the risk of retrograde infection and patient discomfort. Wound drainage has a direct correlation with seroma formation. The loss of protein nutrients and minerals in the serum drained is also a concern with prolonged drainage that can result in healing delays.

The Harmonic™ technology uses ultrasonic energy that allows both cutting and coagulating at the precise point of application. The Harmonic™ has been used since 1992 predominantly in urology and gastro-intestinal surgery (laparoscopic surgery). Significantly reduced serous drainage in a number of general surgery procedures such as superficial and total parotidectomy; thyroidectomy; tonsillectomy; pectoralis major myocutaneous flap dissection; axillary dissection; and lymphadenectomy have been reported with the use Harmonic™.

The Harmonic™ has also been used in parotidectomy and maxillofacial surgery, but its use has been seldom mentioned in the field of plastic and reconstructive surgery. Recent use of the Harmonic™ has shown promise in plastic and reconstructive surgery in dissection of the pectoralis major myocutaneous flap and total body lifts.

Comparisons: The Harmonic™ vs. electrocautery in abdominolipectomy.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this clinical research study must fulfill all of the following criteria:

* Elected to undergo a full abdominoplasty procedure for aesthetics or post-obesity reasons
* Able to comprehend and sign the study informed consent form
* Able to return for all study mandated postoperative visits (3-4 days after the removal of drains, as well as 15 ± 2 days, and 30 ± 5 days after surgery); and
* Be greater than or equal to 18 years of age.

Exclusion Criteria:

Subjects with any of the following criteria are not eligible to participate in this clinical research study:

* Current smoker
* Current use of steroids
* Diabetes Mellitus
* Need of lipocontouring, other than complementary liposuction of the flanks
* Need of a full body lift (belt lipectomy)
* Need of concomitant surgical procedures via the abdominal flap (other than hernia repair, rectus plication, or liposuction of the flanks) or procedures in which the wound drainage would interconnect with the abdominal wound.
* Presence of ventral or umbilical hernia requiring repair with the use of prosthetic material (e.g., mesh)
* Morbid obesity (BMI ≥ 40)
* At risk for ischemia due to presence of obstruction of the arterial blood supply or inadequate blood flow
* Presence of midline scars that could limit flap advancement that are not limited to the infraumbilical region so they can be completely excised
* Right, left, or bilateral upper quadrant scars, (e.g., previous laparotomy via sub costal incision)
* Heart disease
* History of thromboembolic disease
* Current diagnosis or history of any disease that would impair healing process
* Current diagnosis or history of immune system disorders
* History of bleeding disorders
* Presence of uncontrolled hypertension
* Pregnant or lactating
* Being treated with anticoagulants including aspirin within 7 days prior to surgery (a washout period of 7 days will be required); or
* Participation in any other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Total volume (mL) from the time of drain placement to time of drain removal. | from the time of drain placement to time of drain removal

SECONDARY OUTCOMES:
Total number of hours from drain placement to drain removal | from drain placement to drain removal

CONTACTS AND LOCATIONS:
Overall Officials: Drik F Richter, M.D., Principal Investigator — Leiter der Abteilung fuer Plastische Chirurgie
Locations (5):
- United States (2):
  - Iowa City Plastic Surgery, Coralville, Iowa
  - University of Cincinnati, Cincinnati, Ohio
- Centro Zimman de Cirugia Plastica, Buenos Aires, Argentina
- Abteilung für Plastische und Ästhetische Chirurgie, Wesseling, Germany
- Centro Medico Dalinde, Mexico City, Mexico